CLINICAL TRIAL: NCT04948892
Title: Presence of the Father in the Operating Room During Hyperacute Cesarean Section in General Anesthesia
Brief Title: Presence of the Father During Hyperacute Cesarean Section in General Anesthesia
Status: Completed | Type: Observational
Sponsor: Sygehus Lillebaelt (Other)
Responsible Party: Principal Investigator, Helene Korvenius Nedergaard, MD, PhD, Sygehus Lillebaelt
Other Study IDs: SC210815
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Cesarean Section
Keywords: cesarean section; hyperacute cesarean section; family presence; experience of family presence; general anesthesia
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Father/partner present, Kolding hospital: All father/partners, mothers and hospital staff involved in hyperacute cesarean section category 1 in general anesthesia (obstetrician, anesthesiologist, OR-nurse, midwife, anesthetic nurse, pediatrician) in Kolding Hospital, where the father is present in the OR during the cesarean section category 1
  Interventions: Other: Prescence of the father during cesarean section in general anesthesia
- Father/partner not present, Aabenraa hospital: All father/partners and mothers involved in hyperacute cesarean section category 1 in general anesthesia in Aabenraa hospital, where the father is not present in the OR during the cesarean sectio category 1.
  All relevant hospital staff, who sometimes participates in cesarean sectio category 1 (obstetrician, anesthesiologist, OR-nurse, midwife, anesthetic nurse, pediatrician) will be asked to fill in a questionnaire on their thoughts and opinions on having the father/partner present during hyperacute cesarean sectio category 1.

INTERVENTIONS:
Other: Prescence of the father during cesarean section in general anesthesia — The father is now present in the OR during cesarean section category 1, instead of waiting outside
  Groups: Father/partner present, Kolding hospital

SUMMARY:
This study concerns cesarean sections, category 1, meaning those cases where the life of mother and/or fetus is in immedeate danger and the child must be delivered within 15 minutes from activating the cesarean section team. In most hospitals in Denmark, these cesarean sections are most often performed in general anesthesia and the mother is endotracheally intubated.

Previously in these situations, as the mother was rushed from the Labour Ward to the operation room (OR), her spouse/partner, would be placed outside the operating room (OR), and would stay there until the child had been delivered.

In Lillebaelt Hospital, Kolding, Denmark, the newborn-resuscitation table is placed inside the OR. The father would most often be allowed to enter the OR when the child was delivered and placed on the resuscitation table (no matter the status of the child).

However, during spring 2021, Lillebaelt Hospital Kolding updated the policy regarding the handling of the father/partner during cesarean section category 1. Now the father/partner is present in the OR during the whole procedure, including induction of general aesthesia, endotracheal intubation, performance of the cesarean section (drapings are positioned so that the father cannot see the operation field) and potential resuscitation efforts of the newborn.

In another hospital in the same region (Region of Southern Denmark), Aabenraa Hospital, the father is not present in the OR during the cesarean section. He waits in the labour ward.

The investigators therefore wish to investigate how the cesarean section category 1 is experienced by: the father/partner; the mother; the obstetrician; the anestesiologist; the midwife; the OR nurse; the anesthetic nurse, both in Kolding where the father/partner is present in the OR, and in Aabenraa, where the father/partner is not present in the OR during the cesarean sectio.

ELIGIBILITY:
Inclusion Criteria:

* cesarean section category 1

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All mothers and father/partners who experiences a cesarean section category 1 in Kolding Hospital, Denmark.
  All mothers and father/partners who experiences a cesarean section category 1 in Aabenraa Hospital, Denmark
  Hospital staff (obstetricians, anesthesiologists, pediatricians, midwifes, OR-nurses, anesthetic nurses) in Kolding and Aabenraa hospital, who participate in cesarean sectio category 1.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Father/partners experience | 1-2 days after the cesarean section combined with assessment of change from baseline in father/partners experience at 3 months after the cesarean sectio
  Father/partners experience of being present or not in the OR during the hyperacute cesarean section category 1, described by questionnaire, semi-structured interview and PTSD-screening

SECONDARY OUTCOMES:
Mothers experience | 1-2 days after the cesarean section
  Mothers experience of the father/partner being present or not in the OR during the hyperacute cesarean section category 1, described quantitatively with possibility for qualitative components
Surgeons (obstetricians) experience | Up to 2 weeks after the cesarean section
  Surgeons experience of the father/partner being present or not in the OR during the hyperacute cesarean section category 1, described quantitatively with possibility for qualitative components
Anesthesiologists experience | Up to 2 weeks after the cesarean section
  Anesthesiologists experience of the father/partner being present or not in the OR during the hyperacute cesarean section category 1, described quantitatively with possibility for qualitative components
Midwifes experience | Up to 2 weeks after the cesarean section
  Midwifes experience of the father/partner being present or not in the OR during the acute cesarean section category 1, described quantitatively with possibility for qualitative components
OR nurses experience | Up to 2 weeks after the cesarean section
  OR nurses experience of the father being present or not in the OR during the hyperacute cesarean section category 1, described quantitatively with possibility for qualitative components
Anesthetic nurses experience | Up to 2 weeks after the cesarean section
  Anesthetic nurses experience of the father/partner being present or not in the OR during the hyperacute cesarean section category 1, described quantitatively with possibility for qualitative components
Pediatricians experience | Up to 2 weeks after the cesarean section
  Pediatricians experience of the father/partner being present or not in the OR during the hyperacute cesarean section category 1, described quantitatively with possibility for qualitative components

OTHER OUTCOMES:
Obstetric complications | Up to 1 week after the cesarean section
  Perforation of bladder or bowel, bleeding > 1000 ml, infection, need for transfusion
Anesthetic complications | During cesarean section
  Esophageal intubation, difficult airway management
Neonatal complications | During cesarean section
  Low APGAR-score, need for resuscitation, need for intubation, need for transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Hanne I Jensen, Professor, Study Chair — University Hospital of Southern Denmark, Kolding
Locations (2):
- Denmark (2):
  - Aabenraa Hospital, Aabenraa
  - Helene K. Nedergaard, Kolding

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT04948892/SAP_000.pdf